CLINICAL TRIAL: NCT04831294
Title: Effects of Cannabidiol (CBD) on the Brain
Acronym: CBD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Auburn University (Other)
Collaborators: Folium Biosciences (Unknown); FutureCeuticals (Unknown)
Responsible Party: Principal Investigator, Jennifer L. Robinson, Ph.D., Professor, Auburn University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: 20-107 MR 2003
Record Dates: First submitted 2021-04-01; First posted 2021-04-05 (Actual); Last update posted 2023-08-16 (Actual); Status verified 2023-08

CONDITIONS: CBD; Fear; Inhibition
Keywords: cannabidiol; placebo; rct; clinical trial
MeSH Terms: conditions — Inhibition, Psychological | interventions — Cannabidiol

STUDY DESIGN:
Intervention Model Description: Single-site, randomized, placebo-controlled, cross-over, within-subjects design.
  Study sessions are 72 hours apart. Visits included pre-post assessments following ingestion of either placebo or CBD.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Investigators and participants are blind to material assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cannabidiol (CBD) (Experimental): A tincture containing 125mg broad spectrum CBD oil (6.7%), 24mg sunflower lecithin (1.3%), 56mg peppermint oil (3.0%), and 1661mg hempseed oil (89.0%) will be administered orally. Participants will place the liquid in their mouth for 45 seconds before swallowing it.
  Interventions: Drug: Cannabidiol; Drug: Placebo
- Placebo (Placebo Comparator): A tincture containing 149mg sunflower lecithin (8.0%), 56mg peppermint oil (3.0%), 1661mg hempseed oil (89.0%) will be administered orally. Participants will place the liquid in their mouth for 45 seconds before swallowing it.
  Interventions: Drug: Cannabidiol; Drug: Placebo

INTERVENTIONS:
Drug: Cannabidiol — Administered orally. Participants will place the liquid in their mouth for 45 seconds before swallowing it.
  Other Names: CBD
Drug: Placebo — Administered orally. Participants will place the liquid in their mouth for 45 seconds before swallowing it.

SUMMARY:
Cannabidiol (CBD) is a phytocannabinoid that is one of 113 identified cannabinoids in the cannabis plant. It is derived from the hemp plant, and may treat conditions like pain, insomnia, and anxiety. CBD is a critical component of medical marijuana and does not cause the "high" typically associated with cannabis. According to the World Health Organization, CBD has shown no evidence of abuse or dependence potential. However, to the investigator's knowledge, there have not been many acute clinical studies to characterize the effects of CBD in the brain. Despite the rapid influx in CBD readily available to the public, very little is known about such effects. Some studies have shown alterations in resting state connectivity, while others have described changes in specific regions of the brain, or in networks associated with various cognitive functions. For example, CBD has been shown to increase fronto-striatal connectivity and reduce mediotemporal-prefrontal connectivity, suggesting that CBD may affect brain regions involved in salience processing. Unfortunately, few studies have examined CBD in isolation. Additionally, several studies have suggested that CBD may have a neuroprotective effect when it comes to individuals at high risk for psychiatric conditions. In this study, the investigators propose an acute administration, double-blind, placebo-controlled study in which 100% THC-free CBD will be compared to placebo (https://foliumbiosciences.com/). To the investigator's knowledge, the acute effects of this specific product have not been tested. Specifically, the investigators will examine: 1) the neurometabolic and neurophysiological effects of CBD compared to placebo and 2) the behavioral effects of CBD on measures of working memory and response inhibition. Participants will be recruited to take encapsulated, THC-free CBD provided by Folium Biosciences, in which they will have a pre- and post-ingestion scan. Each participant will have a 72-hour washout period after which they will be asked to come back for a placebo scan (however, the order will be counterbalanced so that equal numbers of participants will receive placebo/supplement and supplement/placebo). Individuals will be randomized into the supplementation group, as well as the order.

ELIGIBILITY:
Inclusion Criteria:

1. right-handed
2. between 21-50 years of age
3. no current diagnosis of psychiatric or neurological conditions
4. no history of heart disease or stroke
5. generally healthy
6. pass a screening test for the MR environment

Exclusion Criteria:

1. contraindications to the MR environment
2. use of psychotropic or neurological medication
3. history of heart disease or stroke
4. diabetes or other metabolic conditions
5. self-reported high blood pressure
6. history of concussions
7. any diagnosed psychiatric or neurological condition
8. have consumed alcohol in the 24-hour period prior to a scan
9. consumed pain relievers in the 12-hours prior to a scan
10. consumed food or drinks (except water) and/or nicotine/caffeine an hour prior to any scanning
11. have used or take THC/CBD
12. exercised within an hour of a scan

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2021-07-15 (Actual); Primary Completion 2022-05-15 (Actual); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Behavioral Measures - Change in Go/NoGo Reaction Time | Collected pre-drug, post-drug, pre-placebo, and post-placebo; through study completion (4 time points over a 72 hour period)
  Response/reaction time for each stimuli will be recorded in ms using E-Prime. Reaction times will be calculated for correct and incorrect trials separately.
Behavioral Measures - Change in N-back Reaction Time | Collected pre-drug, post-drug, pre-placebo, and post-placebo; through study completion (4 time points over a 72 hour period)
  Response/reaction time for each stimuli will be recorded in ms using E-Prime. Reaction times will be calculated for correct and incorrect trials separately; and for each level of n-back, separately.
Behavioral Measures - Change in Go/No-Go Accuracy | Collected pre-drug, post-drug, pre-placebo, and post-placebo; through study completion (4 time points over a 72 hour period)
  Accuracy will be determined as the number of trials correct, and errors will be classified as errors of omission or commission.
Behavioral Measures - Change in N-back Accuracy | Collected pre-drug, post-drug, pre-placebo, and post-placebo; through study completion (4 time points over a 72 hour period)
  Accuracy will be determined as the number of trials correct.
Change in Concentration of Neurometabolites | Collected pre-drug, post-drug, pre-placebo, and post-placebo; through study completion (4 time points over a 72 hour period)
  Magnetic resonance spectroscopy (MRS) measurements pre/post ingestion. The following are measured: glutamate, glutamine, gamma-aminobutyric acid, N-acetylaspartate, choline, creatine, glutathione, myo-inositol, aspartate, taurine, and lactate. LCModel software performed automatic quantification of in vivo proton MR spectra by analyzing spectra as a linear combination of model spectra from sequence-specific simulations. Water-suppressed spectra were eddy current corrected and quantified using the unsuppressed water signal. Cramer-Rao lower bounds were used as a measure of fit with CRLB > 50% rejected from further analysis. Metabolite concentrations were CSF-corrected, and quantified (in ppm).
Changes in Functional Connectivity | Collected pre-drug, post-drug, pre-placebo, and post-placebo; through study completion (4 time points over a 72 hour period)
  Blood-oxygen-level-dependent signal changes will be collected via functional magnetic resonance imaging (fMRI). We will assess pre- and post-drug/placebo connectivity changes across the whole-brain using standard preprocessing procedure (fmriprep) and the 'conn' connectivity toolbox.
Blood Oxygen Level Dependent (BOLD) Changes | Collected pre-drug, post-drug, pre-placebo, and post-placebo; through study completion (4 time points over a 72 hour period)
  Functional magnetic resonance imaging blood-oxygen-level-dependent signal changes across tasks, and during resting state
BOLD - Change in Threat Response to Subliminal Emotion Stimuli | Collected pre-drug, post-drug, pre-placebo, and post-placebo; through study completion (4 time points over a 72 hour period)
  Responses to emotional face stimuli will be measured as a function of blood-oxygen-level-dependent signal change during emotion versus neutral condition in predefined regions of interest including the amygdala, anterior cingulate cortex, and superior temporal sulcus.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer L Robinson, Ph.D., Principal Investigator — Auburn University
Locations (1):
- Auburn University MRI Research Center, Auburn, Alabama, United States

IPD SHARING:
Plan to Share IPD: Undecided
Our consent form does include an optional item for participants to indicate whether or not they would be agreeable to their data being shared.

REFERENCES:
- [Background] Grimm O, Loffler M, Kamping S, Hartmann A, Rohleder C, Leweke M, Flor H. Probing the endocannabinoid system in healthy volunteers: Cannabidiol alters fronto-striatal resting-state connectivity. Eur Neuropsychopharmacol. 2018 Jul;28(7):841-849. doi: 10.1016/j.euroneuro.2018.04.004. Epub 2018 Jun 7. PMID 29887287
- [Background] Wall MB, Pope R, Freeman TP, Kowalczyk OS, Demetriou L, Mokrysz C, Hindocha C, Lawn W, Bloomfield MA, Freeman AM, Feilding A, Nutt D, Curran HV. Dissociable effects of cannabis with and without cannabidiol on the human brain's resting-state functional connectivity. J Psychopharmacol. 2019 Jul;33(7):822-830. doi: 10.1177/0269881119841568. Epub 2019 Apr 23. PMID 31013455
- [Background] Beale C, Broyd SJ, Chye Y, Suo C, Schira M, Galettis P, Martin JH, Yucel M, Solowij N. Prolonged Cannabidiol Treatment Effects on Hippocampal Subfield Volumes in Current Cannabis Users. Cannabis Cannabinoid Res. 2018 Apr 1;3(1):94-107. doi: 10.1089/can.2017.0047. eCollection 2018. PMID 29682609
- [Background] Wilson R, Bossong MG, Appiah-Kusi E, Petros N, Brammer M, Perez J, Allen P, McGuire P, Bhattacharyya S. Cannabidiol attenuates insular dysfunction during motivational salience processing in subjects at clinical high risk for psychosis. Transl Psychiatry. 2019 Aug 22;9(1):203. doi: 10.1038/s41398-019-0534-2. PMID 31439831
- [Background] O'Neill A, Wilson R, Blest-Hopley G, Annibale L, Colizzi M, Brammer M, Giampietro V, Bhattacharyya S. Normalization of mediotemporal and prefrontal activity, and mediotemporal-striatal connectivity, may underlie antipsychotic effects of cannabidiol in psychosis. Psychol Med. 2021 Mar;51(4):596-606. doi: 10.1017/S0033291719003519. Epub 2020 Jan 29. PMID 31994476
- [Background] Bhattacharyya S, Falkenberg I, Martin-Santos R, Atakan Z, Crippa JA, Giampietro V, Brammer M, McGuire P. Cannabinoid modulation of functional connectivity within regions processing attentional salience. Neuropsychopharmacology. 2015 May;40(6):1343-52. doi: 10.1038/npp.2014.258. Epub 2014 Sep 23. PMID 25249057
- [Background] Borgwardt SJ, Allen P, Bhattacharyya S, Fusar-Poli P, Crippa JA, Seal ML, Fraccaro V, Atakan Z, Martin-Santos R, O'Carroll C, Rubia K, McGuire PK. Neural basis of Delta-9-tetrahydrocannabinol and cannabidiol: effects during response inhibition. Biol Psychiatry. 2008 Dec 1;64(11):966-73. doi: 10.1016/j.biopsych.2008.05.011. Epub 2008 Jun 27. PMID 18589404
- [Background] Allendorfer JB, Nenert R, Bebin EM, Gaston TE, Grayson LE, Hernando KA, Houston JT, Hansen B, Szaflarski JP. fMRI study of cannabidiol-induced changes in attention control in treatment-resistant epilepsy. Epilepsy Behav. 2019 Jul;96:114-121. doi: 10.1016/j.yebeh.2019.04.008. Epub 2019 May 24. PMID 31129526
- [Background] Bhattacharyya S, Wilson R, Appiah-Kusi E, O'Neill A, Brammer M, Perez J, Murray R, Allen P, Bossong MG, McGuire P. Effect of Cannabidiol on Medial Temporal, Midbrain, and Striatal Dysfunction in People at Clinical High Risk of Psychosis: A Randomized Clinical Trial. JAMA Psychiatry. 2018 Nov 1;75(11):1107-1117. doi: 10.1001/jamapsychiatry.2018.2309. PMID 30167644
- [Background] Pretzsch CM, Voinescu B, Mendez MA, Wichers R, Ajram L, Ivin G, Heasman M, Williams S, Murphy DG, Daly E, McAlonan GM. The effect of cannabidiol (CBD) on low-frequency activity and functional connectivity in the brain of adults with and without autism spectrum disorder (ASD). J Psychopharmacol. 2019 Sep;33(9):1141-1148. doi: 10.1177/0269881119858306. Epub 2019 Jun 25. PMID 31237191
- [Background] Hermann D, Sartorius A, Welzel H, Walter S, Skopp G, Ende G, Mann K. Dorsolateral prefrontal cortex N-acetylaspartate/total creatine (NAA/tCr) loss in male recreational cannabis users. Biol Psychiatry. 2007 Jun 1;61(11):1281-9. doi: 10.1016/j.biopsych.2006.08.027. Epub 2007 Jan 17. PMID 17239356
- [Background] Fusar-Poli P, Crippa JA, Bhattacharyya S, Borgwardt SJ, Allen P, Martin-Santos R, Seal M, Surguladze SA, O'Carrol C, Atakan Z, Zuardi AW, McGuire PK. Distinct effects of delta9-tetrahydrocannabinol and cannabidiol on neural activation during emotional processing. Arch Gen Psychiatry. 2009 Jan;66(1):95-105. doi: 10.1001/archgenpsychiatry.2008.519. PMID 19124693
- [Background] Bhattacharyya S, Morrison PD, Fusar-Poli P, Martin-Santos R, Borgwardt S, Winton-Brown T, Nosarti C, O' Carroll CM, Seal M, Allen P, Mehta MA, Stone JM, Tunstall N, Giampietro V, Kapur S, Murray RM, Zuardi AW, Crippa JA, Atakan Z, McGuire PK. Opposite effects of delta-9-tetrahydrocannabinol and cannabidiol on human brain function and psychopathology. Neuropsychopharmacology. 2010 Feb;35(3):764-74. doi: 10.1038/npp.2009.184. Epub 2009 Nov 18. PMID 19924114